CLINICAL TRIAL: NCT02098811
Title: Evaluation of the Safety and Efficacy of a Non-Invasive Disruption of Fat and Skin Tightening Using 1064nm and 940nm Wavelengths
Brief Title: Evaluation of the Safety and Precursors of Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: CYN13-NIF-JD-04
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Subcutaneous Fat
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1064nm laser Treatment Before Abdominoplasty (Experimental): Patient will be treated with 1064nm Laser prior to abdominoplasty
  Interventions: Device: 1064nm Laser
- 940nm Laser Treatment Before Abdominoplasty (Experimental): Patient will be treated with 940nm Laser prior to abdominoplasty
  Interventions: Device: 940nm Laser

INTERVENTIONS:
Device: 1064nm Laser — Patient will be treated with 1064nm Laser prior to abdominoplasty
  Arms: 1064nm laser Treatment Before Abdominoplasty
Device: 940nm Laser — Patient will be treated with 940nm Laser prior to abdominoplasty
  Arms: 940nm Laser Treatment Before Abdominoplasty

SUMMARY:
The purpose of this study is to evaluate and compare the safety and pre-cursors of efficacy of a non-invasive 1064nm laser and 940nm diode, for the disruption of subcutaneous adipose tissue and skin tightening.

DETAILED DESCRIPTION:
The purpose of the biopsies is to assess if the device causes an inflammatory response in the abdominoplasty tissue that will be excised.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking subjects between ages of 20-55 years of age presenting excess abdominal tissue (fat and skin), are candidates for an abdominoplasty procedure and are willing to allow the use of this device on their skin
* Subjects (Group 2 and 3) who will allow the excess skin removed as part of the abdominoplasty to be sent for laboratory analysis
* Understand and accept the obligation associated with the procedure
* Subjects with Fitzpatrick skin types I to VI.
* Subjects (Group 2 and 3) who are willing to consent to participate in the study will be asked to undergo treatment, elasticity and ultrasound measurements, as outlined for each group and defined in section 6.0.
* Subjects must agree to maintain the same diet and exercise regime throughout the study

Exclusion Criteria:

* Any previous liposuction/lipo-sculpture or any type of procedure in the abdominal area in the past 6 months
* A history of allergic reactions to medications or anesthesia required for the procedure
* A history of thrombophlebitis
* A history of acute infections
* A history of heart failure
* Received or is anticipated to receive antiplatelets, anticoagulants, thrombolytics, vitamin E or anti-inflammatories within 2 weeks pre treatment
* Intolerance to anesthesia or medications to be prescribed before or after the procedure.
* Any medical condition, that, in the investigator's opinion would interfere with the patient's participation in the study
* Taking medications that are photosensitive
* A history of keloid formation
* A study subject must not be pregnant or have been pregnant in the last 3 months
* The physician has the right to make determination of eligibility as he/she determines based on the standard of care

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Biopsy of Tissue Sample as a Measure of Effectiveness | 6 months post treatment
  Biopsy of treated area will be obtained up to 6 months post treatment and will be histologically assessed for changes in adipocytes, collagen and surrounding tissue to determine effectiveness of device
Ultrasound Measurement to Evaluate Reduction of Fat | 6 months post treatment
  Ultrasound of the treatment area will be performed and evaluated in comparison to the baseline results to determine reduction of fat

SECONDARY OUTCOMES:
High Frequency Ultrasound to Measure Skin Elasticity and Thickness | 6 months post last treatment
  High frequency ultrasound of the treatment area will be performed and evaluated in comparison to baseline results to measure changes in skin elasticity and skin thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Patric Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Aesthetic Pavilion, Staten Island, New York, United States